CLINICAL TRIAL: NCT05175235
Title: Nivolumab and Pembrolizumab Dose Optimisation in Solid Tumours With CURATE.AI Platform and Sequential ctDNA Measurements
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: The N.1 Institute for Health (N.1) (Other); Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/00334-Immunotherapy
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor
Keywords: personalized oncology; personalized dose selection; immunotherapy; dose optimisation; Cancer; Artificial Intelligence; CURATE.AI; Nivolumab; Sequential ctDNA; Chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, one-arm, prospective pilot study of participants diagnosed with solid tumours. The participants will be enrolled for the duration of their treatment with Nivolumab. At 12-month mark, the decision on the patient engagement with the study will be made by the principal investigator in consultation with the study sponsors and treating physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CURATE.AI (Experimental): Participants will undergo two treatment periods: selection period and CURATE.AI modulation period. During the selection period, baseline ctDNA measurements and CT scans will be performed. Subsequently, participants will receive Standard of Care (SOC) doses of nivolumab/pembrolizumab and have their ctDNA measured at the end of the third cycle together with other SOC monitoring.
  After the first ctDNA measurement and CT scan, selected patients who responded to treatment through both ctDNA and CT scan may continue into the CURATE.AI modulation period. Non-responders will receive SOC doses of nivolumab/pembrolizumab for 2 cycles before having their ctDNA measured and CT scan at the end of the 2 cycles. Subsequent responders through both ctDNA and CT scans may then continue into the CURATE.AI modulation period.
  Only the dose of nivolumab/pembrolizumab will be modulated with CURATE.AI, based on measurements of the response marker (ctDNA).
  Interventions: Device: CURATE.AI; Drug: Nivolumab, Pembrolizumab

INTERVENTIONS:
Device: CURATE.AI — Efficacy and toxicity measurements at the end of each two-/three- week dosing cycle, together with an information on given drugs and their doses, and other patient data, will be used by CURATE.AI to recommend the dose of nivolumab/pembrolizumab for the next cycle. The clinical investigators will decide whether or not to administer or prescribe the dose recommendation from CURATE.AI.
Drug: Nivolumab, Pembrolizumab — Treatment with the selected regimen will take up to a maximum duration of 12 months, in two-/three- week cycles. CURATE.AI dose recommendations will be generated before each chemotherapy cycle; fixed throughout the cycle; Maximum total cumulative dose per cycle of nNivolumab/pembrolizumab in the predetermined safety range is set at 100% of standard starting dose (i.e. , 240 mg/m2 once every 2 weeks for single agent Nivolumab and 200 mg/m2 once every 3 weeks for single agent Pembrolizumab). Minimum total cumulative dose per cycle of nivolumab/pembrolizumab in the predetermined safety range is set at 30% of the standard starting dose (i.e. 8072 mg/m2 once every 2 weeks for single agent Nivolumab and 60 mg/m2 once every 3 weeks for single agent Pembrolizumab). Subject-specific dosing range may alter those numbers to suit the specific circumstances of the subject, thus giving the subject specific safe dosing range.

SUMMARY:
CURATE.AI - a small data, AI-derived technology platform - allows personalised guidance of an individual's dose modulations based only on that individual's data. Additionally, CURATE.AI is mechanism-independent, and dynamically adapts to changes experienced by the subject, providing dynamic dose optimisation throughout the duration of the subject's treatment. This study aims to demonstrate the feasibility of applying CURATE.AI in standard of care settings for treatment of solid tumours with Nivolumab. An additional objective is to explore sequential ctDNA measurements as a response marker collected at a higher frequency of probing, with modulated doses.

DETAILED DESCRIPTION:
The first stage of the trial aims to identify patients who are responsive to the given treatment, determined from both SOC - radiology via criteria such as RECIST/immune-related RECIST (irRECIST) as well as the intended response marker for CURATE.AI. These patients will then proceed with the second stage of the trial.

The second stage of the trial aims to obtain a personalised CURATE.AI profile for each participant, based on their phenotypic response to a set of drug doses. The doses will be recommended by the CURATE.AI team, when relevant to the clinical decision-making process. For participants who started on the selected therapy prior to their engagement with the study, the previously recorded data, limited to: administered doses, corresponding phenotypic responses and treatment-related toxicities (optional) may be included in the CURATE.AI process. Once an actionable profile is obtained, dose recommendations are based on the profile and aimed to treat the participant.

Since there are no prior clinical trials using CURATE.AI in participant treated with combinational or single-agent immunotherapy with drugs such as nivolumab or pembrolizumab, this trial will comprise of participants diagnosed with the main tumour types: non-small cell lung cancer (NSCLC), gastric cancer (GC), hepatocellular carcinoma (HCC) or nasopharyngeal carcinoma (NPC), or other eligible tumours undergoing or planned for palliative-intent immune-oncology combinational or single-agent therapy with nivolumab/ pembrolizumab.

Nivolumab and Pembrolizumab are an immune checkpoint inhibitors and a novel therapeutic treatment modalities recently approved by the FDA and are becoming the standard of care treatment for a range of oncological indications, including NSCLC, GC, HCC and NPC. However, they are associated with significant semi-annual costs - approximately $140,000 per patient in the United States. In light of the evidence supporting dose personalization and dose reduction in immune-oncology treatments, patients may stand to benefit from CURATE.AI's personalized dose optimisation in maximizing clinical outcomes at reduced costs. Together with the increasing adoption of circulating tumour DNA (ctDNA) as an effective response marker for tumour burden in NSCLC, GC, HCC and NPC, CURATE.AI is ideally suited for pairing these findings with healthcare economics research towards the development of novel healthcare workflows integrating AI and serial measurements of ctDNA response to sustain the scalable implementation of N-of-1 dosing optimisation in cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 21 years of age
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
3. Patients must meet the following clinical laboratory criteria within 21 days of starting treatment:

   1. Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3
   2. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN of ≤ 5 ULN if involvement of the liver.
   3. Calculated creatinine clearance ≥ 30 mL/min or creatinine < 1.5 x ULN.
4. Main tumour types: Non-small cell lung cancer (NSCLC), gastric cancer (GC), hepatocellular carcinoma (HCC) and nasopharyngeal carcinoma (NPC) or other metastatic solid tumours not for curative intent therapy;
5. Treatment with combinational immunotherapy or single-agent nivolumab/pembrolizumab. If patients have already started treatment on this regimen, they may still be eligible to enrol, provided they fulfil all other criteria and approval is sought by PI and Sponsor.
6. Eligible for treatment combinational immunotherapy or single-agent nivolumab /pembrolizumab based on co-investigator's assessment of fitness for immunotherapy (e.g. not on high dose corticosteroid therapy or uncontrolled auto-immune disorder)

Exclusion Criteria:

1. Patients who are lactating or pregnant.
2. Patients with clinically significant hypersensitivity to one or more of the selected regimen's constituent drug(s)
3. Contraindication to any of the required concomitant drugs or supportive treatments.
4. Any clinically significant medical disease or psychiatric condition that, in the co-investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.
5. Major surgery within 28 days prior to start of the treatment,
6. Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischaemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 4 months prior to informed consent obtained.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants in whom we successfully apply CURATE.AI profile. | up to 12 months
  CURATE.AI applicability: Percentage of participants in whom we successfully apply CURATE.AI profile. Based on percentages, outcomes will be classified as Green (>70%) / Yellow (10-70%) / Red (<10%).
  A decision on whether we "successfully apply" the CURATE.AI profile requires expert judgement and cannot be made based on a purely numerical process. The expert panel will consider the following factors with careful regard for the individual circumstances of each participant:
  Error/variance (biological/analytical) is sufficiently small to allow accurate predictions Profile can be generated sufficiently early for the participant to potentially benefit; Dose-dependent relationship is observed; Profile is actionable (i.e. fulfils the clinical investigator's pre-specified safety requirements); Systemic changes in the participant which require profile recalibration are rare or readily assimilated into the CURATE.AI algorithm

SECONDARY OUTCOMES:
Patient adherence | Up to 12 months
  Percentage of participants who always adhered to the prescribed dose whenever they took their medication, as measured by the standardised pharmacovigilance protocol. Based on percentages, outcomes will be classified as Green (>90%) / Yellow (10-90%) / Red (<10%).
Timely delivery of CURATE.AI recommendations to the clinician | Up to 12 months
  Percentage of CURATE.AI recommendations provided in time for the next chemotherapy cycle, across all participants and cycles. Based on percentages, outcomes will be classified as Green (100%) / Yellow (10-99%) / Red (<10%).
CURATE.AI relevance | Up to 12 months
  Percentage of dosing events across all participants and cycles in which CURATE.AI recommendation is considered in the clinical decision-making process. Based on percentages, outcomes will be classified as Green (100%) / Yellow (10-99%) / Red (<10%).
Physician adherence | Up to 12 months
  Percentage of CURATE.AI recommended doses that were used by the clinical investigator. Based on percentages, outcomes will be classified as Green (>70%) / Yellow (10-70%) / Red (<10%).
Clinically significant dose changes | Up to 12 months
  Percentage of participants in whom the CURATE.AI-guided cumulative dose is substantially (≥10%) different from the projected standard-of-care cumulative dose. Based on percentages, outcomes will be classified as Green (>20%) / Yellow (1-20%) / Red (0%).

OTHER OUTCOMES:
Percentage of trial participants with clinical progressive disease | Up to 12 months
  CT scans for radiological assessment will be performed according to standard of care, usually after every 2 to 3 cycles of chemotherapy Percentage of trial participants with clinical progressive disease(which is defined as the clinical investigator deeming that the patient will not benefit any further from the chemotherapy regimen and considering stopping it) at the time of the first radiological assessment performed as per standard-of-care.
Temporal variation in response marker (ctDNA) level from baseline to trial conclusion. | Up to 12 months
  Mandatory blood draws for the measurement of response marker(s)as per standard of care. Additional blood draws solely for the purposes of the trial for measurements of response markers(s) Tumour marker measurements at higher frequency will be analysed to inform about temporal dynamics of tumour response to modulated dosing.
Maximal reduction in response marker (ctDNA) level measured as part of baseline investigations | Up to 12 months
  For CURATE.AI profile generation, a minimum of 3 dose levels and corresponding response marker readouts are needed for the modulated drug. After obtaining the first response marker readout a set of potential doses to pick from will be recommended by the CURATE.AI team with calibration-intent, based on the mathematical requirements of the method.
Toxicity derived from the use of CURATE.AI | Up to 12 months
  Percentage of trial participants with clinically relevant toxicities of grades 3-4 based on CTCAE version 4.0.
ctDNA analysis | Up to 12 months
  Data collection and explorative analysis of ctDNA as:
  1. As response marker in serial measurements at given clinical context and after modulated dosing in comparison to radiology (via criteria such as RECIST/immune related RECIST (irRECIST) for monitoring treatment response dynamics in the immuno-oncology;
  2. As a potential input for CURATE.AI

CONTACTS AND LOCATIONS:
Overall Officials: Raghav Sundar, Principal Investigator — NUH
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin JC, Wang WY, Chen KY, Wei YH, Liang WM, Jan JS, Jiang RS. Quantification of plasma Epstein-Barr virus DNA in patients with advanced nasopharyngeal carcinoma. N Engl J Med. 2004 Jun 10;350(24):2461-70. doi: 10.1056/NEJMoa032260. PMID 15190138
- [Result] Kazandjian D, Suzman DL, Blumenthal G, Mushti S, He K, Libeg M, Keegan P, Pazdur R. FDA Approval Summary: Nivolumab for the Treatment of Metastatic Non-Small Cell Lung Cancer With Progression On or After Platinum-Based Chemotherapy. Oncologist. 2016 May;21(5):634-42. doi: 10.1634/theoncologist.2015-0507. Epub 2016 Mar 16. PMID 26984449
- [Result] Evan TH, Jenny Z, Eun-Jeong K, Grace H, Shailender B, Sunil AR. Economic analysis of alternative pembrolizumab and nivolumab dosing strategies at an academic cancer centre. JCO 2019; 37(15): 6504-6504. doi: 10.1200/JCO.2019.37.15_suppl.6504
- [Result] Yoo SH, Keam B, Kim M, Kim SH, Kim YJ, Kim TM, Kim DW, Lee JS, Heo DS. Low-dose nivolumab can be effective in non-small cell lung cancer: alternative option for financial toxicity. ESMO Open. 2018 Jul 25;3(5):e000332. doi: 10.1136/esmoopen-2018-000332. eCollection 2018. PMID 30094065
- [Result] Low JL, Huang Y, Sooi K, Ang Y, Chan ZY, Spencer K, Jeyasekharan AD, Sundar R, Goh BC, Soo R, Yong WP. Low-dose pembrolizumab in the treatment of advanced non-small cell lung cancer. Int J Cancer. 2021 Jul 1;149(1):169-176. doi: 10.1002/ijc.33534. Epub 2021 Mar 6. PMID 33634869